CLINICAL TRIAL: NCT04030260
Title: Regorafenib and PD-1 Antibody in Combination With Radiotherapy With or Without SBRT in Patients With pMMR/MSS and Previously Treated Metastatic Colorectal Cancer
Brief Title: Regorafenib and PD-1 Antibody in Combination With Radiotherapy for pMMR/MSS Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-16
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer Metastatic; MSS
MeSH Terms: interventions — regorafenib; Radiotherapy; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib and PD-1 antibody in Combination with Radiotherapy (Experimental)
  Interventions: Drug: Regorafenib and PD-1 antibody in Combination with Radiotherapy; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Regorafenib and PD-1 antibody in Combination with Radiotherapy — Regorafenib will be given 3 weeks on/1 week off (80 mg od po.) and PD-1 antibody
  Other Names: Regorafenib; PD-1 antibody
Radiation: Radiation therapy — Radiation therapy is believed to increase the likelihood of response of immunotherapy

SUMMARY:
REGONIVO is a Phase Ib study to explore the efficacy and safety of regorafenib in combination with nivolumab in the treatment of gastric cancer and colorectal cancer with MSS. The study enrolled 50 patients with advanced disease, including 25 cases of gastric cancer, 25 cases of colorectal cancer, except for one case of colorectal cancer with MSI-H, and others were MSS type. The results of the study showed that patients with colorectal cancer had an objective response rate (ORR) of 36% and a progression-free survival (PFS) of 6.3 months.

Based on the preliminary results of the REGONIVO study, the aim of this phase 2 study is to explore the safety and efficacy of regorafenib and PD-1 antibody with or without radiotherapy in previously treated metastatic colorectal cancer patients with pMMR/MSS.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
* Subjects with metastatic colorectal cancer(CRC) (Stage IV).
* Subjects must have failed at least two lines of prior treatment.
* Tumor tissues were identified as mismatch repair-proficient (pMMR) by immunohistochemistry (IHC) method or microsatellite stability (MSS) by polymerase chain reaction (PCR).
* Progression during or within 3 months following the last administration of approved standard therapies which must include a fluoropyrimidine, oxaliplatin and irinotecan.

  * Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy.
  * Subjects who progress more than 6 months after completion of oxaliplatin containing adjuvant treatment must be retreated with oxaliplatin-based therapy to be eligible.
  * Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed into the study.
  * Subjects may have received prior treatment with Avastin (bevacizumab) and/or Erbitux (cetuximab)/Vectibix (panitumumab) (if KRAS WT)
* Metastatic CRC subjects must have measurable or non measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 1.
* Life expectancy of at least 3 months.
* Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol.

Exclusion Criteria:

* Prior treatment with Regorafenib.
* Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T-lymphocyte-associated Protein 4, CTLA-4) antibody or other drug/antibody that acts on T cell costimulation or checkpoint pathways.
* Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to randomization.
* Cardiological disease including Congestive heart failure, Unstable angina, Myocardial infarction, Cardiac arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension. (Systolic blood pressure 150 mmHg or diastolic pressure 90 mmHg despite optimal medical management).
* Pleural effusion or ascites that causes respiratory compromise.
* Arterial or venous thrombotic or embolic events.
* Any history of or currently known brain metastases.
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 4 week.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-07-19 (Estimated)

PRIMARY OUTCOMES:
The progression-free survival (PFS) rates at 6 months | 2 year
  The PFS is defined as the time from the start of treatment to the date of first documented PD or death as a result of any cause, whichever occurred first. When a patient was alive and without progression, PFS was censored at the date of the last disease assessment. The PFS rates at 6 months was estimated from Kaplan-Meier curves.

SECONDARY OUTCOMES:
The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR). | 2 year
Overall Survival (OS) | 2 year
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Disease Control Rate (DCR) | 2 year
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)
Safety variables will be summarized using descriptive statistics based on adverse events collection | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No